CLINICAL TRIAL: NCT04731571
Title: Toward High Fidelity Adaptive Radiotherapy in the Thorax
Status: Completed | Type: Observational
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Joshua Kim, Medical Physicist, Henry Ford Health System
Other Study IDs: HighFidelityART
Record Dates: First submitted 2021-01-26; First posted 2021-02-01 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Radiotherapy: Patients with locally advanced non-small cell lung cancer previously treated with definitive chemoradiotherapy

SUMMARY:
Daily adaptive radiotherapy with individualized planning margins for thoracic and pelvic cancer patients will increase the potential of reducing dose to OARs, thereby reducing treatment-related toxicities and ultimately providing these patients with a better quality of life. Thus, the overarching objective of this work is to develop a CBCT-guided adaptive workflow and to measure the benefits to patients of the adaptive treatment paradigm utilizing patient reported outcomes in a first-of-kind study.

DETAILED DESCRIPTION:
1. To individualize the planning margins used for treatment, we will assess the impact of the different uncertainties on patient-specific planning margins. We determine the dosimetric uncertainties for patients during planning and delivery through the daily adaptive process. In so doing, we will determine the relationship between the dose distributions and the associated treatment outcomes.
2. To perform retrospective clinical studies using patient data, we determine the relationship between dosimetry from plans developed using the optimized patient-specific margins (plans from (1) that are robust to uncertainties) and retrospective, clinical outcomes. This data will be used to inform daily adaptation and plan quality criteria for a prospective clinical protocol.
3. To develop (with our clinical collaborators) a first-of-kind study to measure the efficacy of daily adaptive treatment with individualized planning margins, using clinical and quality of life (patient reported) outcomes, and to compare these against the conventional treatment approach, where a single treatment plan with population-based treatment margins is utilized for all treatment fractions.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed non-small cell lung cancer patients
* Locally advanced

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with unresectable, locally advanced non-small cell lung cancer
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-02-05 (Actual); Primary Completion 2024-10-22 (Actual); Study Completion 2025-02-27 (Actual)

PRIMARY OUTCOMES:
The number of patients with treatment-related Grade 3 or higher adverse cardiac events as defined by the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE v5.0) at 2 years | through study completion, an average of 2 years
  A set of treatment planning strategies were designed and retrospectively implemented for locally advanced, non-small cell lung cancer (NSCLC) patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Health, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim JP, Dewalt J, Feldman A, Adil K, Movsas B, Chetty IJ. Feasibility of radical cardiac-sparing, treatment planning strategies for patients with locally advanced, non-small cell lung cancer. J Appl Clin Med Phys. 2022 Dec;23(12):e13784. doi: 10.1002/acm2.13784. Epub 2022 Oct 13. PMID 36237114
- [Background] Yan D, Georg D. Adaptive radiation therapy. Z Med Phys. 2018 Aug;28(3):173-174. doi: 10.1016/j.zemedi.2018.03.001. Epub 2018 Mar 27. No abstract available. PMID 29602589
- [Background] Zhong H, Siddiqui SM, Movsas B, Chetty IJ. Evaluation of adaptive treatment planning for patients with non-small cell lung cancer. Phys Med Biol. 2017 Jun 7;62(11):4346-4360. doi: 10.1088/1361-6560/aa586f. Epub 2017 Jan 10. PMID 28072395
- [Background] Herschtal A, Te Marvelde L, Mengersen K, Foroudi F, Eade T, Pham D, Caine H, Kron T. Sparing healthy tissue and increasing tumor dose using bayesian modeling of geometric uncertainties for planning target volume personalization. Int J Radiat Oncol Biol Phys. 2015 Jun 1;92(2):446-52. doi: 10.1016/j.ijrobp.2015.01.034. Epub 2015 Apr 3. PMID 25847606
- [Background] Dial C, Weiss E, Siebers JV, Hugo GD. Benefits of adaptive radiation therapy in lung cancer as a function of replanning frequency. Med Phys. 2016 Apr;43(4):1787. doi: 10.1118/1.4943564. PMID 27036576